CLINICAL TRIAL: NCT05369039
Title: The Potential Therapeutic Effect of Roflumilust (a Selective Phosphodiesterase 4inhibitor) on Chronic Rhinosinusitis With Nasal Polyposis.
Brief Title: Roflumilust in Chronic Rhinosinusitis With Nasal Polyposis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmad Mahmoud Hamdan, Principal Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2022 ENT
Record Dates: First submitted 2022-03-03; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Chronic Sinusitis
Keywords: Roflumilust; Chronic Sinusitis with nasal polyposis; Phosphodiesterase inhibitor
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to the patient's group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Case Group (Experimental): The case group will receive a 10 days course of Roflumilust in a dose of 500 mg once daily.
  Interventions: Drug: Roflumilust
- Control group (Active Comparator): The Control group will receive a 10 days course of systemic steroids in the form of oral prednisolone in a dose of 40 mg per day.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Roflumilust — A selective phosphodiesterase 4 Inhibitor
  Arms: Case Group
Drug: Prednisolone — Systemic corticosteroid
  Arms: Control group

SUMMARY:
The current study will be a pilot study for a randomized controlled trial conducted on 60 patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine after approval of the institutional review board and taking informed written consent from every patient before participation in the study. The patients of this study will be randomly and equally distributed among case and control groups to compare the effect of Roflumilust administration with the effect of systemic and local corticosteroids on patients with chronic rhinosinusitis with nasal polyposis

DETAILED DESCRIPTION:
The current study will be a pilot study for a randomized controlled trial conducted on 60 patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine after approval of the institutional review board and taking informed written consent from every patient before participation in the study. The patients of this study will be randomly and equally distributed among case and control groups.

To be included in the study, patients should be more than 18 years old, have chronic rhinosinusitis with nasal polyposis, and have no history of systemic steroid administration over the last three months. History of previous nasal surgery, underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases), and hypersensitivity to Roflumilust were the exclusion criteria for this study.

Patients of the study will be randomly and equally distributed between case and control groups using block randomization methods using 4 blocks each comprising 4 patients with 6 patterns for every block one of which was selected randomly using random numbers generated by Excel program. The case group will receive a 10 days course of Roflumilust in a dose of 500 mg once daily. The Control group will receive a 10 days course of systemic steroids in the form of oral prednisolone in a dose of 40 mg per day.

Assessment protocol:

Patients of the study will be assessed before and at the end of the treatment protocol with history taking to define the inclusion and exclusion criteria and to assess the burden of nasal symptoms using SNOT-22 scale. Endoscopic examination of the nasal cavity will be performed to confirm the presence of bilateral nasal polyposis and to assess the degree of nasal polyposis using the Lund Kennedy score. Serum IL17 and periostin will be assessed using ELISA technique before and after treatment to assess the anti-inflammatory effects of the drug.

Outcome measures:

Primary outcome measures will include a comparison between the pre and post treatment values of SNOT-22 and Lund Kennedy scores, serum IL17, and serum priostin in both case and control groups. Another outcome measure will be the comparison between the case and control groups regarding the posttreatment and posttreatment values of the previous indices. Secondary outcome measures will include an assessment of the side effects of Roflumilust among the case group.

ELIGIBILITY:
Inclusion Criteria:

* chronic rhinosinusitis with nasal polyposis,
* No history of systemic steroid administration over the last three months

Exclusion Criteria:

* History of previous nasal surgery,
* Underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases),
* Hypersensitivity to Roflumilust

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between pretreatment and posttreatment SNOT-22 score in both groups | 2 weeks after start of treatment
  Post-treatment SNOT-22 scores will be compared with pretreatment scores in both groups
Comparison between pretreatment and posttreatment Lund Kennedy scores in both groups | Two weeks after start of treatment
  Post-treatment Lund Kennedy scores will be compared with pretreatment scores in both groups
Comparison between pretreatment and posttreatment Serum periostin levels in both groups | Two weeks after start of treatment
  Post-treatment Serum periostin level in pg/ml will be compared with pretreatment levels in both group
Comparison between case and control groups regarding SNOT 22 score | Two weeks after start of treatment
  Case and control groups are compared regarding post-treatment SNOT-22 score
Comparison between case and control groups regarding Lund Kennedy score | Two weeks after start of treatment
  Case and control groups are compared regarding post-treatment Lund Kennedy score
Comparison between case and control groups regarding serum periostin level | Two weeks after start of treatment
  Case and control groups are compared regarding post-treatment serum periostin level in pg/ml

SECONDARY OUTCOMES:
Assessment of the side effects of Roflumilust | Two weeks after start of treatment
  The side effects of Roflumilust will be assessed among the case group

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data is available on request from the authors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the study
Access Criteria: After approval of the authors on request

REFERENCES:
- [Background] Hulse KE, Stevens WW, Tan BK, Schleimer RP. Pathogenesis of nasal polyposis. Clin Exp Allergy. 2015 Feb;45(2):328-46. doi: 10.1111/cea.12472. PMID 25482020
- [Background] Ryu G, Bae JS, Kim JH, Kim EH, Lyu L, Chung YJ, Mo JH. Role of IL-17A in Chronic Rhinosinusitis With Nasal Polyp. Allergy Asthma Immunol Res. 2020 May;12(3):507-522. doi: 10.4168/aair.2020.12.3.507. PMID 32141263
- [Background] Maxfield AZ, Landegger LD, Brook CD, Lehmann AE, Campbell AP, Bergmark RW, Stankovic KM, Metson R. Periostin as a Biomarker for Nasal Polyps in Chronic Rhinosinusitis. Otolaryngol Head Neck Surg. 2018 Jan;158(1):181-186. doi: 10.1177/0194599817737967. Epub 2017 Oct 17. PMID 29040053
- [Background] Janosova V, Calkovsky V, Pedan H, Behanova E, Hajtman A, Calkovska A. Phosphodiesterase 4 Inhibitors in Allergic Rhinitis/Rhinosinusitis. Front Pharmacol. 2020 Jul 22;11:1135. doi: 10.3389/fphar.2020.01135. eCollection 2020. PMID 32792957
- [Background] Inagaki N, Miura T, Daikoku M, Nagai H, Koda A. Inhibitory effects of beta-adrenergic stimulants on increased vascular permeability caused by passive cutaneous anaphylaxis, allergic mediators, and mediator releasers in rats. Pharmacology. 1989;39(1):19-27. doi: 10.1159/000138567. PMID 2479953